CLINICAL TRIAL: NCT04172441
Title: A Randomized Trial in 2 Parts: Double-Blind, Placebo-Controlled, Crossover Part 1 and Open-label Part 2, Evaluating the Efficacy and Safety of Dasiglucagon for the Treatment of Children With Congenital Hyperinsulinism
Brief Title: Trial Evaluating Efficacy and Safety of Dasiglucagon in Children With Congenital Hyperinsulinism
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Zealand Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZP4207-17103; 2017-004545-24 (EudraCT Number)
Record Dates: First submitted 2019-11-18; First posted 2019-11-21 (Actual); Results first posted 2025-03-14 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Congenital Hyperinsulinism
MeSH Terms: conditions — Congenital Hyperinsulinism | interventions — dasiglucagon

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- dasiglucagon first then placebo (Experimental): 48 hours of dasiglucagon subcutaneous (sc) infusion starting at 10 µg/hour with crossover to 48 hours placebo sc infusion (part 1) followed by 21 days of dasiglucagon sc infusion (part 2).
  Interventions: Drug: dasiglucagon; Drug: Placebo
- placebo first then dasiglucagon (Experimental): 48 hours of placebo sc infusion with crossover to 48 hours dasiglucagon sc infusion starting at 10 µg/hour (part 1) followed by 21 days of dasiglucagon sc infusion (part 2).
  Interventions: Drug: dasiglucagon; Drug: Placebo

INTERVENTIONS:
Drug: dasiglucagon — Glucagon analogue
  Other Names: ZP4207
Drug: Placebo — Placebo for dasiglucagon

SUMMARY:
The objective of the trial is to evaluate the efficacy of dasiglucagon in reducing glucose requirements in children with persistent congenital hyperinsulinism (CHI) requiring continuous intravenous (IV) glucose administration to prevent/manage hypoglycemia.

ELIGIBILITY:
Inclusion Criteria:

* CHI diagnosis established based on the following:

  1. Hyperinsulinemia: plasma insulin above the limit of detection of the assay documented during an event of hypoglycemia, and/or
  2. Hypofattyacidemia: plasma free fatty acid <1.7 mmol/L, and/or
  3. Hypoketonemia: Beta-hydroxybutyrate <1.8 mmol/L, and/or
  4. Glycemic response: an increase in plasma glucose (PG) of >30 mg/dL (1.7 mmol/L) after 1 mg IV or intramuscular (IM) glucagon administration
* Male or female, age ≥7 days and <12 months at screening
* Body weight of ≥2.0 kg (4.4 lbs.)
* Continuous IV glucose requirement to prevent hypoglycemia

Exclusion Criteria:

* Is suspected of having a transient form of CHI (e.g., transient hyperinsulinism due to maternal diabetes or perinatal stress)
* Was born preterm below 34 weeks of gestational age
* Presence of hypertension or hypotension, including circulatory instability requiring supportive medication or presence of pheochromocytoma
* Known or suspected presence of severe brain damage
* Evidence of metabolic, endocrine, or syndromic causes of hypoglycemia not due to hyperinsulinism
* Use of systemic corticosteroids, e.g., hydrocortisone >20 mg/m^2 body surface area or equivalent within 5 days before screening
* Prior use of lanreotide, sirolimus (mechanistic target of rapamycin [mTOR] inhibitors), anti-inflammatory biological agents, or other immune modulating agents. Prior use of octreotide is allowed after a minimum of 48 hour washout before randomization.
* Any clinically significant abnormality identified on echocardiogram that in the opinion of the investigator would affect the subject's ability to participate in the trial
* Any recognized clotting or bleeding disorder
* The use of prescription or non-prescription medications known to cause QT prolongation

Ages: 7 Days to 364 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2020-06-19 (Actual); Primary Completion 2022-02-17 (Actual); Study Completion 2022-03-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jelena Ivkovic, MD, Study Director — Zealand Pharma
Locations (6):
- United States (2):
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Cook Children's Medical Center, Fort Worth, Texas
- Germany (2):
  - University Children's Hospital, Düsseldorf
  - University Hospital, Magdeburg, Magdeburg
- Hadassah Medical Center, Jerusalem, Israel
- Manchester University NHS Foundation Trust, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Dasiglucagon, Then Placebo: Patients were treated with dasiglucagon for 48 hours in Part 1-1, then placebo for 48 hours in Part 1-2, and then dasiglucagon for 21 days in Part 2
- Placebo, Then Dasiglucagon: Patients were treated with placebo for 48 hours in Part 1-1, then dasiglucagon for 48 hours in Part 1-2, and then dasiglucagon for 21 days in Part 2
Period: Part 1-1: First Intervention (48 Hours)
Arm/Group | Dasiglucagon, Then Placebo | Placebo, Then Dasiglucagon
Started | 7 | 5
Completed | 7 | 5
Not Completed | 0 | 0
Period: Part 1-2: Second Intervention (48 Hours)
Arm/Group | Dasiglucagon, Then Placebo | Placebo, Then Dasiglucagon
Started | 7 | 5
Completed | 7 | 5
Not Completed | 0 | 0
Period: Part 2: Open Label Dasiglucagon
Arm/Group | Dasiglucagon, Then Placebo | Placebo, Then Dasiglucagon
Started | 7 | 5
Completed Treatment | 7 | 4 (1 participant discontinued treatment during Part 2 of the study.)
Completed | 7 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants Who Received Treatment: All participants who received treatment
Arm/Group | All Participants Who Received Treatment
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 12
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: Days] | 71.25 (84.976)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 2
  Race: White | 8
  Race: Other | 2
Region of Enrollment [Number; unit: participants]
  United States | 8
  United Kingdom | 3
  Germany | 1
Gastrostomy/nasogastric tube [Count of Participants; unit: Participants]
  Gastrostomy | 2
  Nasogastric tube | 7
  None | 3

OUTCOME MEASURES:

1. Primary Outcome: Mean Intravenous Glucose Infusion Rate
Description: Mean intravenous (IV) glucose infusion rate (GIR) in the last 12 hours of each treatment period during Part 1, the crossover part of the trial (dasiglucagon or placebo administration).
Time Frame: Hours 36-48 after initiation of trial drug (Part 1)
Measure: Mean (Standard Deviation); unit: mg/kg/minute
Groups:
- Dasiglucagon: All patients treated with dasiglucagon in Part 1
- Placebo: All patients treated with placebo in Part 1
Arm/Group | Dasiglucagon | Placebo
Number analyzed (Participants) | 12 | 12
mg/kg/minute | 4.33 (4.922) | 9.51 (5.655)
Statistical Analysis 1: Comparison: Dasiglucagon vs Placebo; Null hypothesis: weighted mean IV GIR in the last 12 hours of treatment with dasiglucagon = weighted mean IV GIR in the last 12 hours of treatment with placebo; Test type: Superiority; p = 0.0037, Mixed Models Analysis; A mixed model was used, with treatment and period as fixed effects and patient as random effect; Difference in LS means = -5.21, 95% CI 2-sided [-8.29 to -2.13] — The comparison was in the direction of dasiglucagon minus placebo

2. Secondary Outcome: Carbohydrates Administered
Description: Total amount (g) of carbohydrates administered during the crossover part of the trial (dasiglucagon or placebo administration) per day.
Time Frame: 0 to 48 hours after initiation of trial drug
Measure: Mean (Standard Deviation); unit: g/day
Arm/Group | Dasiglucagon | Placebo
Number analyzed (Participants) | 12 | 12
g/day | 106.7 (53.72) | 139.1 (57.35)
Statistical Analysis 1: Comparison: Dasiglucagon vs Placebo; Null hypothesis: Total amount of carbohydrates administered (regardless of route) per day in patients treated with dasiglucagon = total amount of carbohydrates administered (regardless of route) per day in patients treated with placebo; Test type: Superiority; p = 0.0238, Mixed Models Analysis; A mixed model was used, with treatment and period as fixed effects and patient as random effect; Difference in LS means = -30.93, 95% CI 2-sided [-56.80 to -5.05] — The comparison was in the direction of dasiglucagon minus placebo

3. Secondary Outcome: Mean Intravenous Glucose Infusion Rate
Description: Mean IV GIR for each 48-hour treatment period during Part 1, the crossover part of the trial (dasiglucagon or placebo administration).
Time Frame: 48 hours after initiation of trial drug (Part 1)
Measure: Mean (Standard Deviation); unit: mg/kg/minute
Arm/Group | Dasiglucagon | Placebo
Number analyzed (Participants) | 12 | 12
mg/kg/minute | 6.9 (5.91) | 10.4 (5.31)

4. Secondary Outcome: Mean Intravenous Glucose Infusion Rate Below 10 mg/kg/Minute
Description: Mean IV GIR below 10 mg/kg/minute in the last 12 hours of each treatment period during Part 1, the crossover part of the trial (dasiglucagon or placebo administration) (yes/no)
Time Frame: Hours 36-48 after initiation of trial drug (Part 1)
Measure: Count of Participants; unit: Participants
Arm/Group | Dasiglucagon | Placebo
Number analyzed (Participants) | 12 | 12
Participants
  Mean IV GIR below 10 mg/kg/min in the last 12 hours of each treatment period during Part 1?: yes | 9 | 6
  Mean IV GIR below 10 mg/kg/min in the last 12 hours of each treatment period during Part 1?: no | 3 | 6

5. Secondary Outcome: Time to Complete Weaning Off Intravenous Glucose
Description: Time in days to complete weaning off IV glucose administration during Part 2, defined as the first point in time when the patient had been off IV glucose administration for at least 12 hours.
Time Frame: Days 5 to 25 (Part 2)
Measure: Median (95% Confidence Interval); unit: days
Groups:
- Dasiglucagon (Part 2): All patients treated with dasiglucagon in Part 2
Arm/Group | Dasiglucagon (Part 2)
Number analyzed (Participants) | 12
days | 5.8 [1.0 to 7.9]

6. Secondary Outcome: Hypoglycemia Event Rate in Part 2
Description: Hypoglycemia event rate, defined as number of hypoglycemic events when PG was <70 mg/dL (or 3.9 mmol/L), as detected by self-monitored plasma glucose.
Time Frame: Days 5 to 25
Population: Self-monitored plasma glucose episodes were set to missing after pancreatectomy; 2 patients had near-total or partial pancreatectomies during Part 2 of the study.
Measure: Median (Full Range); unit: episodes per week
Arm/Group | Dasiglucagon (Part 2)
Number analyzed (Participants) | 12
episodes per week
  Week 1 (Days 5 to 11) | 8.50 [0.0 to 29.0]
  Week 2 (Days 12 to 18): number analyzed (Participants) | 11
  Week 2 (Days 12 to 18) | 6.0 [0.0 to 37.3]
  Week 3 (Days 19 to 25): number analyzed (Participants) | 10
  Week 3 (Days 19 to 25) | 3.79 [0.0 to 15.2]
  Weeks 1 to 3 (Days 5 to 25) | 6.04 [1.7 to 33.2]

7. Secondary Outcome: Clinically Significant Hypoglycemia Events in Part 2
Description: Clinically significant hypoglycemia event rate, defined as number of events when PG was <54 mg/dL (3.0 mmol/L), as detected by self-monitored plasma glucose.
Time Frame: Days 5 to 25
Population: as for outcome 6
Measure: Median (Full Range); unit: episodes per week
Arm/Group | Dasiglucagon (Part 2)
Number analyzed (Participants) | 12
episodes per week
  Week 1 (Days 5 to 11) | 1.67 [0.0 to 11.0]
  Week 2 (Days 12 to 18): number analyzed (Participants) | 11
  Week 2 (Days 12 to 18) | 1.00 [0.0 to 16.3]
  Week 3 (Days 19 to 25): number analyzed (Participants) | 10
  Week 3 (Days 19 to 25) | 2.92 [0.0 to 4.0]
  Weeks 1 to 3 (Days 5 to 25) | 1.67 [0.3 to 13.7]

8. Secondary Outcome: Time to Actual Hospital Discharge
Description: Time in days to actual hospital discharge defined as the time from first exposure to the study drug in Part 2 to discharge from hospital.
Time Frame: Days 5 to 25
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Dasiglucagon (Part 2)
Number analyzed (Participants) | 12
days | NA [11.7 to NA] — A median value and upper limit of the 95% confidence interval were not calculable due to an insufficient number of patients being discharged from hospital.

9. Secondary Outcome: Time to Pancreatic Surgery
Description: Time (days) to pancreatic surgery (sub-total or total pancreatectomy with a cutoff of ≥95%).
Time Frame: Days 5 to 25
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Dasiglucagon (Part 2)
Number analyzed (Participants) | 12
days | NA [NA to NA] — The median value and 95% confidence interval were not calculable due to an insufficient number of patients undergoing sub-total or total pancreatectomy with a cutoff of ≥95%.

10. Secondary Outcome: Carbohydrates Administered
Description: Total amount (g) of carbohydrates administered (regardless of the route) per day.
Time Frame: Days 5 to 25
Population: Carbohydrates amount administered was set to missing after pancreatectomy; 2 patients had near-total or partial pancreatectomies during Part 2 of the study.
Measure: Median (Full Range); unit: g/day
Arm/Group | Dasiglucagon (Part 2)
Number analyzed (Participants) | 12
g/day
  Week 1 (Days 5 to 11) | 91.03 [57.6 to 190.8]
  Week 2 (Days 12 to 18): number analyzed (Participants) | 11
  Week 2 (Days 12 to 18) | 75.09 [29.8 to 218.3]
  Week 3 (Days 19 to 25): number analyzed (Participants) | 10
  Week 3 (Days 19 to 25) | 80.73 [0.0 to 222.1]
  Weeks 1 to 3 (Days 5 to 25) | 87.37 [39.5 to 195.9]

11. Secondary Outcome: Carbohydrates Administered Intravenously
Description: Amount (g) of carbohydrates administered via IV glucose infusion or bolus or total parenteral nutrition. This secondary endpoint was intended to account only for carbohydrates administered via IV glucose infusion or bolus. It was not possible to differentiate between carbohydrates administered via IV glucose infusion or bolus and carbohydrates administered as being, or not being, part of total parenteral nutrition from the collected data. This endpoint was expanded to include both.
Time Frame: Days 5 to 25
Population: as for outcome 10
Measure: Median (Full Range); unit: g/day
Arm/Group | Dasiglucagon (Part 2)
Number analyzed (Participants) | 12
g/day
  Week 1 (Days 5 to 11) | 41.35 [3.6 to 118.8]
  Week 2 (Days 12 to 18): number analyzed (Participants) | 11
  Week 2 (Days 12 to 18) | 2.12 [0.0 to 82.2]
  Week 3 (Days 19 to 25): number analyzed (Participants) | 10
  Week 3 (Days 19 to 25) | 0.35 [0.0 to 119.0]
  Weeks 1 to 3 (Days 5 to 25) | 22.60 [1.2 to 88.5]

12. Secondary Outcome: Carbohydrates Administered Parenterally
Description: Amount (g) of carbohydrates administered as part of total parenteral nutrition.
Time Frame: Days 5 to 25
Population: It was not possible to differentiate between carbohydrates administered via IV glucose infusion or bolus and carbohydrates administered as being, or not being, part of total parenteral nutrition because some of the carbohydrates that were given as a part of parenteral nutrition were also reported as carbohydrates administered intravenously. All available results regarding administration of carbohydrates are presented in outcome measure 11.
Arm/Group | Dasiglucagon (Part 2)
Number analyzed (Participants) | 0

13. Secondary Outcome: Carbohydrates Administered Orally
Description: Amount (g) of carbohydrates administered via oral route.
Time Frame: Days 5 to 25
Population: as for outcome 10
Measure: Median (Full Range); unit: g/day
Arm/Group | Dasiglucagon (Part 2)
Number analyzed (Participants) | 12
g/day
  Week 1 (Days 5 to 11) | 19.57 [0.0 to 67.5]
  Week 2 (Days 12 to 18): number analyzed (Participants) | 11
  Week 2 (Days 12 to 18) | 0.37 [0.0 to 88.9]
  Week 3 (Days 19 to 25): number analyzed (Participants) | 10
  Week 3 (Days 19 to 25) | 0.23 [0.0 to 53.8]
  Weeks 1 to 3 (Days 5 to 25) | 13.38 [0.0 to 63.4]

14. Secondary Outcome: Carbohydrates Administered Via Gastric Feed
Description: Amount (g) of carbohydrates administered via nasogastric tube or gastrostomy.
Time Frame: Days 5 to 25
Population: as for outcome 10
Measure: Median (Full Range); unit: g/day
Arm/Group | Dasiglucagon (Part 2)
Number analyzed (Participants) | 12
g/day
  Week 1 (Days 5 to 11) | 34.43 [0.0 to 88.7]
  Week 2 (Days 12 to 18): number analyzed (Participants) | 11
  Week 2 (Days 12 to 18) | 52.87 [9.0 to 92.8]
  Week 3 (Days 19 to 25): number analyzed (Participants) | 10
  Week 3 (Days 19 to 25) | 57.90 [0.0 to 76.1]
  Weeks 1 to 3 (Days 5 to 25) | 43.96 [0.0 to 85.0]

15. Secondary Outcome: Time in Range in Part 2
Description: Percent time in range (PG between 70 to 180 mg/dL [3.9-10.0 mmol/L]) as measured by continuous glucose monitoring.
Time Frame: Days 5 to 25
Population: Data were not available from all patients during all weeks.
Measure: Median (Full Range); unit: percent time
Arm/Group | Dasiglucagon (Part 2)
Number analyzed (Participants) | 12
percent time
  Week 1 (Days 5 to 11): number analyzed (Participants) | 11
  Week 1 (Days 5 to 11) | 86.69 [34.5 to 94.3]
  Week 2 (Days 12 to 18): number analyzed (Participants) | 10
  Week 2 (Days 12 to 18) | 87.87 [51.0 to 95.9]
  Week 3 (Days 19 to 25): number analyzed (Participants) | 10
  Week 3 (Days 19 to 25) | 91.42 [36.3 to 100.0]
  Weeks 1 to 3 (Days 5 to 25) | 88.35 [42.5 to 100.0]

16. Secondary Outcome: Time in Hypoglycemia in Part 2
Description: Percent time in hypoglycemia (when PG was <70 mg/dL [or 3.9 mmol/L]) as measured by continuous glucose monitoring.
Time Frame: Days 5 to 25
Population: Data were not available from all patients during all weeks.
Measure: Median (Full Range); unit: percent time
Arm/Group | Dasiglucagon (Part 2)
Number analyzed (Participants) | 12
percent time
  Week 1 (Days 5 to 11): number analyzed (Participants) | 11
  Week 1 (Days 5 to 11) | 7.20 [1.0 to 24.5]
  Week 2 (Days 12 to 18): number analyzed (Participants) | 10
  Week 2 (Days 12 to 18) | 8.82 [0.6 to 49.0]
  Week 3 (Days 19 to 25): number analyzed (Participants) | 10
  Week 3 (Days 19 to 25) | 5.73 [0.0 to 22.1]
  Weeks 1 to 3 (Days 5 to 25) | 6.67 [0.0 to 30.0]

17. Secondary Outcome: Time in Clinically Significant Hypoglycemia in Part 2
Description: Percent time in clinically significant hypoglycemia (when PG was <54 mg/dL [or 3.0 mmol/L]) as measured by continuous glucose monitoring.
Time Frame: Days 5 to 25
Population: Data were not available from all patients during all weeks.
Measure: Median (Full Range); unit: percent time
Arm/Group | Dasiglucagon (Part 2)
Number analyzed (Participants) | 12
percent time
  Week 1 (Days 5 to 11): number analyzed (Participants) | 11
  Week 1 (Days 5 to 11) | 2.07 [0.2 to 6.0]
  Week 2 (Days 12 to 18): number analyzed (Participants) | 10
  Week 2 (Days 12 to 18) | 2.20 [0.0 to 20.4]
  Week 3 (Days 19 to 25): number analyzed (Participants) | 10
  Week 3 (Days 19 to 25) | 0.88 [0.0 to 6.8]
  Weeks 1 to 3 (Days 5 to 25) | 1.75 [0.0 to 9.2]

18. Secondary Outcome: Hypoglycemia Episodes in Part 2
Description: Rate of hypoglycemia episodes, defined as number of episodes per week when PG was <70 mg/dL (3.9 mmol/L) for 15 minutes or more, as measured by continuous glucose monitoring.
Time Frame: Days 5 to 25
Population: Data were not available from all patients during all weeks.
Measure: Median (Full Range); unit: episodes per week
Arm/Group | Dasiglucagon (Part 2)
Number analyzed (Participants) | 12
episodes per week
  Week 1 (Days 5 to 11): number analyzed (Participants) | 11
  Week 1 (Days 5 to 11) | 25.00 [3.0 to 58.0]
  Week 2 (Days 12 to 18): number analyzed (Participants) | 10
  Week 2 (Days 12 to 18) | 26.50 [3.0 to 74.7]
  Week 3 (Days 19 to 25): number analyzed (Participants) | 10
  Week 3 (Days 19 to 25) | 18.63 [0.0 to 58.3]
  Weeks 1 to 3 (Days 5 to 25) | 18.54 [0.0 to 66.3]

19. Secondary Outcome: Clinically Significant Hypoglycemia Episodes in Part 2
Description: Rate of clinically significant hypoglycemia episodes, defined as number of episodes per week when was <54 mg/dL (3.0 mmol/L) for 15 minutes or more, as measured by continuous glucose monitoring.
Time Frame: Days 5 to 25
Population: Data were not available from all patients during all weeks.
Measure: Median (Full Range); unit: episodes per week
Arm/Group | Dasiglucagon (Part 2)
Number analyzed (Participants) | 12
episodes per week
  Week 1 (Days 5 to 11): number analyzed (Participants) | 11
  Week 1 (Days 5 to 11) | 5.00 [1.0 to 23.0]
  Week 2 (Days 12 to 18): number analyzed (Participants) | 10
  Week 2 (Days 12 to 18) | 8.50 [0.0 to 46.7]
  Week 3 (Days 19 to 25): number analyzed (Participants) | 10
  Week 3 (Days 19 to 25) | 2.67 [0.0 to 18.7]
  Weeks 1 to 3 (Days 5 to 25) | 5.00 [0.0 to 34.8]

20. Secondary Outcome: Extent of Hypoglycemia in Part 2
Description: Extent of hypoglycemia (defined as the area over the glucose curve [AOCglucose] below 70 mg/dL [3.9 mmol/L]) as measured by continuous glucose monitoring.
Time Frame: Days 5 to 25
Population: Data were not available from all patients during all weeks.
Measure: Median (Full Range); unit: mg/dL/hour
Arm/Group | Dasiglucagon (Part 2)
Number analyzed (Participants) | 12
mg/dL/hour
  Week 1 (Days 5 to 11): number analyzed (Participants) | 11
  Week 1 (Days 5 to 11) | 0.87 [0.1 to 2.7]
  Week 2 (Days 12 to 18): number analyzed (Participants) | 10
  Week 2 (Days 12 to 18) | 0.97 [0.0 to 8.9]
  Week 3 (Days 19 to 25): number analyzed (Participants) | 9
  Week 3 (Days 19 to 25) | 0.59 [0.1 to 2.6]
  Weeks 1 to 3 (Days 5 to 25): number analyzed (Participants) | 11
  Weeks 1 to 3 (Days 5 to 25) | 0.89 [0.1 to 4.3]

21. Secondary Outcome: Extent of Clinically Significant Hypoglycemia in Part 2
Description: Extent of clinically significant hypoglycemia (defined as the area over the glucose curve [AOCglucose] below 54 mg/dL [3.0 mmol/L]) as measured by continuous glucose monitoring, divided by the total duration in hours of continuous glucose monitoring.
Time Frame: Days 5 to 25
Population: Data were not available from all patients during all weeks.
Measure: Median (Full Range); unit: mg/dL/hour
Arm/Group | Dasiglucagon (Part 2)
Number analyzed (Participants) | 12
mg/dL/hour
  Week 1 (Days 5 to 11): number analyzed (Participants) | 11
  Week 1 (Days 5 to 11) | 0.14 [0.0 to 0.4]
  Week 2 (Days 12 to 18): number analyzed (Participants) | 9
  Week 2 (Days 12 to 18) | 0.13 [0.0 to 2.1]
  Week 3 (Days 19 to 25): number analyzed (Participants) | 8
  Week 3 (Days 19 to 25) | 0.12 [0.0 to 0.4]
  Weeks 1 to 3 (Days 5 to 25): number analyzed (Participants) | 11
  Weeks 1 to 3 (Days 5 to 25) | 0.14 [0.0 to 0.8]

22. Secondary Outcome: Time in Hyperglycemia in Part 2
Description: Percent time in hyperglycemia (when PG was >180 mg/dL [10.0 mmol/L]), as measured by continuous glucose monitoring.
Time Frame: Days 5 to 25
Population: Data were not available from all patients from all weeks.
Measure: Median (Full Range); unit: percent time
Arm/Group | Dasiglucagon (Part 2)
Number analyzed (Participants) | 12
percent time
  Week 1 (Days 5 to 11): number analyzed (Participants) | 11
  Week 1 (Days 5 to 11) | 1.74 [0.0 to 64.5]
  Week 2 (Days 12 to 18): number analyzed (Participants) | 10
  Week 2 (Days 12 to 18) | 0.81 [0.0 to 45.0]
  Week 3 (Days 19 to 25): number analyzed (Participants) | 10
  Week 3 (Days 19 to 25) | 0.32 [0.0 to 62.7]
  Weeks 1 to 3 (Days 5 to 25) | 1.48 [0.0 to 56.6]

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are reported here, and were recorded from the time of first administration of study treatment until the end of the posttreatment follow-up period or inclusion in the ZP4207-17106 extension trial (up to 8 weeks, from Day 1 through Day 56).
Description: Note that the reporting groups are not mutually exclusive.
Groups:
- Part 1: Dasiglucagon: Adverse events during administration of dasiglucagon during Part 1 of the study.
- Part 1: Placebo: Adverse events during administration of placebo during Part 1 of the study.
- Part 2: Dasiglucagon: Adverse events during administration of dasiglucagon during Part 2 of the study.
- Parts 1 and 2: Dasiglucagon: Adverse events during administration of dasiglucagon during Parts 1 and 2 of the study.
- Follow-up Period: Adverse events occurring during the Follow-up Period.
Arm/Group | Part 1: Dasiglucagon | Part 1: Placebo | Part 2: Dasiglucagon | Parts 1 and 2: Dasiglucagon | Follow-up Period
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/12 | 0/12 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 1/12 | 1/12 | 0/1
Other Adverse Events (participants affected / at risk) | 3/12 | 7/12 | 10/12 | 10/12 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: Dasiglucagon (N=12) | Part 1: Placebo (N=12) | Part 2: Dasiglucagon (N=12) | Parts 1 and 2: Dasiglucagon (N=12) | Follow-up Period (N=1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: Dasiglucagon (N=12) | Part 1: Placebo (N=12) | Part 2: Dasiglucagon (N=12) | Parts 1 and 2: Dasiglucagon (N=12) | Follow-up Period (N=1)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (2) | 0 (0)
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2) | 3 (3) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (1)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Aspartate Aminotransferase Increased (Investigations) | 1 (1) | 1 (1) | 2 (2) | 2 (3) | 0 (0)
Alanine Aminotransferase Increased (Investigations) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Finger Deformity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash Papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (3) | 3 (3) | 0 (0)
Dermatitis Diaper (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Acne Infantile (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dry Skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Seborrhoeic Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Sensitive Skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (3) | 2 (3) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (4) | 2 (4) | 0 (0)
Acidosis Hyperchloraemic (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Fluid Retention (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hypochloraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 0 (0)
Face Oedema (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Medical Device Site Reaction (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Thrombophlebitis Superficial (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 3 (4) | 3 (4) | 0 (0)
Normocytic Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Device Related Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Eye Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Fungal Skin Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 0 (0)
Oral Candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Parainfluenzae Virus Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Rash Pustular (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dry Eye (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Procedural Pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Haemangioma Of Liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Device Occlusion (Product Issues) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-06-04): https://cdn.clinicaltrials.gov/large-docs/41/NCT04172441/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-08): https://cdn.clinicaltrials.gov/large-docs/41/NCT04172441/SAP_001.pdf